CLINICAL TRIAL: NCT05091749
Title: Detection of Significant Coronary Artery Disease by Promising Biomarker: A2A Adenosine Receptor (A2AR) Assays
Acronym: ADOCAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-16; 2021-A02200-41 (Other: IDRCB)
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Coronary Syndromes
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic coronary syndromes (Experimental)
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — troponin measurement

SUMMARY:
Transversal, national, multi-center study with progressive recruitment designed to assess the diagnostic accuracy of A2AR expression for the identification of significant obstructive CAD (FFR<0.8) of patients suspected of CCS compared to the gold standard.

1. To assess the diagnostic accuracy of the A2AR profile (i.e. KD/EC50) for identifying myocardial ischemia in patients with suspected CCS compared to the gold standard inducible myocardial ischemia.
2. To determine the best threshold value for A2AR expression for identifying significant obstructive CAD (FFR<0,8) in patients with CCS, and to estimate the diagnostic performances associated with the identified threshold
3. To determine the best threshold value for A2AR profile (i.e. KD/EC50) for identifying myocardial ischemia (See annex 2) in patients with CCS and to estimate the diagnostic performances associated with the identified threshold.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged ≥18 and <90 years old;
* Must not be of child-bearing potential (≥1 year post-menopausal, contraceptive, or surgically sterile);
* Symptoms suggestive of CCS and intermediate PTP (15-85%) according to the Diamond classification (2);
* Undergone at least one stress imaging test (annex 3) or an abnormal coronary Computed Tomography Angiography (CTA) with the recommendation to perform ICA with FFR in all intermediate lesions;
* Non-contributive ECG (resting 18-lead);
* Normal echocardiography with left ventricular ejection fraction (LVEF) >50%;
* Cardiac troponin level <99th percentile;
* Intended for an invasive strategy for CCS;
* Affiliated to or beneficiary of, a social security system;
* Signed written informed consent.

Exclusion Criteria:

Persons referred in articles L.1121-5 to L.1121-8 and L.1122-2 of the Public Health Code:

* Pregnant, parturient or breastfeeding woman
* Person deprived of liberty for judicial or administrative decision
* Person under psychiatric care
* Minor person (non-emancipated)

  * History of CAD or known CAD
  * Suspected acute coronary syndrome (ACS: annex 4)
  * Inability to undergo adenosine testing
  * Allergy to iodinated contrast media
  * Bleeding diathesis
  * Known significant bleeding risk according to physician judgment
  * Severe hepatic failure (ASAT, ALAT>3ULN)
  * Ischemic stroke within 1 month or a history of hemorrhagic stroke
  * Bradycardia
  * Platelet count <100 G/L
  * Hemoglobin <10g/dl
  * Major surgery or trauma within 10 days
  * Life expectancy <1 year
  * Pre-test Probability <15% or >85%
  * History and clinical examination suggesting non-cardiac chest pain
  * Contraindication to coronary angiography
  * Thyroid disorder
  * Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
A 2AR measure | 24 MONTHS
  blood sample

CONTACTS AND LOCATIONS:
Overall Officials: CREMIEUX François, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France